CLINICAL TRIAL: NCT00112307
Title: Pilot Study of Magnetic Resonance Imaging Guided Brachytherapy
Brief Title: Magnetic Resonance Imaging Guided Gynecologic Brachytherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03-201; NCT00165113 (obsolete NCT alias)
Record Dates: First submitted 2005-06-01; First posted 2005-06-02 (Estimated); Last update posted 2009-09-17 (Estimated); Status verified 2009-09

CONDITIONS: Cervix Neoplasms; Uterine Neoplasms; Vaginal Neoplasms; Vulvar Neoplasms
Keywords: MRI; Brachytherapy; Carcinoma; Cervix; Uterus; Vagina; Vulva; Carcinoma of the cervix; Carcinoma of the uterus; Carcinoma of the vagina; Carcinoma of the vulva
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Neoplasms; Vaginal Neoplasms; Vulvar Neoplasms; Carcinoma | interventions — Brachytherapy

INTERVENTIONS:
Procedure: Brachytherapy

SUMMARY:
The primary goal of this pilot study is to assess the feasibility of using magnetic resonance (MR) imaging guidance in the Magnetic Resonance Therapy (MRT) unit at the Brigham and Women's Hospital during the implantation of brachytherapy applicators in patients with gynecologic malignancies. Patients with gynecologic malignancies requiring brachytherapy are currently treated under either fluoroscopic or CT visualization of the brachytherapy applicator. Magnetic resonance imaging has been shown in many studies to provide superior visualization of the cervix, vagina and uterus compared to CT. However no prior study has examined the feasibility of using real-time magnetic resonance imaging to assist in the guidance of gynecologic brachytherapy applicators

DETAILED DESCRIPTION:
The primary endpoint involves the ability of the MRT guided procedure to protect bladder and rectal tissues from inadvertent insertion of the interstitial needles used to deliver brachytherapy. MR images obtained on the MRT unit should provide clear delineation of the bladder and rectum and allow for greater accuracy and avoidance of these normal tissues upon interstitial needle insertion. CT images will be obtained following the insertion of needles using the MRT unit. The procedure will be considered a failure if CT imaging identifies the insertion of needles into the bladder or rectum that was not detected using MR. Secondary endpoints include the ability of MR imaging to accurately reconstruct dosimetric plans and to construct dose volume histograms after the implantation of interstitial needles as well as the ability of MR imaging to accurately determine tumor, bladder and rectal volumes. Secondary endpoints will also include the assessment of acute skin, genitourinary and gastrointestinal toxicities as well as an assessment of tumor progression or recurrence during a 180 day follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Histologic documentation of carcinoma. Carcinoma of the cervix: Stage IIIB, IVA or vaginal recurrence
* Carcinoma of the cervix: Stage IB, IIA, IIB or IIIA with obliteration of the cervical os (tandem and ovoid implant not feasible)
* Carcinoma of the uterus: Stage IIIB (vaginal involvement) or vaginal recurrence
* Carcinoma of the vagina: Stage II, III, IVA or vaginal recurrence
* Carcinoma of the vulva: T3 (vaginal extension) or T4 (inoperable - any N stage), or vaginal recurrence
* MRI and CT of the pelvis within 2 months before registration
* ECOG performance status of < 2
* Age > 18
* Signed informed consent
* No metallic objects or pacemakers in the patient
* Negative pregnancy test for those of child-bearing potential
* Patients who have received prior radiation or chemotherapy may be enrolled on this study.
* Documented complete blood count (CBC) with hematocrit (Hct)>30, absolute neutrophil count (ANC)>500, platelet (Plt) >40

Exclusion Criteria:

* Patients with distant metastasis.
* Baseline studies not obtained.
* Patients who are pregnant or lactating.
* Significant history of cardiovascular disease.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15
Dates: Start 2003-03; Study Completion 2005-10

PRIMARY OUTCOMES:
Insertion of needles into the bladder or rectum

SECONDARY OUTCOMES:
Ability of MR imaging to accurately determine tumor, bladder and rectal volumes
Assessment of acute skin, genitourinary and gastrointestinal toxicities
Assessment of tumor progression or recurrence during a 180 day follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Akila N Viswanathan, MD, MPH, Principal Investigator — BWH/DFCI